CLINICAL TRIAL: NCT04431193
Title: Estimate Serum Oxytocin Pharmacodynamic Range in the Periphery
Brief Title: Estimate Serum Oxytocin PD Range in the Periphery
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study will be replaced by a revised study protocol
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00066130
Record Dates: First submitted 2020-06-05; First posted 2020-06-16 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-05

CONDITIONS: Osteoarthritis, Knee
Keywords: advanced knee arthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Oxytocin infused to maintain serum concentrations of 4, 16, 64, and 256 picogram/millilitre
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Oxytocin 4 picogram/millilitre (Experimental): Oxytocin infused to maintain serum concentration of 4 picogram/millilitre
  Interventions: Drug: Oxytocin
- Oxytocin 16 picogram/millilitre (Experimental): Oxytocin infused to maintain serum concentration of 16 picogram/millilitre
  Interventions: Drug: Oxytocin
- Oxytocin 64 picogram/millilitre (Experimental): Oxytocin infused to maintain serum concentration of 64 picogram/millilitre
  Interventions: Drug: Oxytocin
- Oxytocin 256 picogram/millilitre (Experimental): Oxytocin infused to maintain serum concentration of 256 picogram/millilitre
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — Oxytocin infused to maintain serum concentrations of 4, 16, 64, and 256 picogram/millilitre
  Other Names: Pitocin

SUMMARY:
The main purpose of this study is to define the maximum effect oxytocin (naturally occurring hormone that is made in the brain) has on pain from a 5 minute heat probe applied to the skin and to get an estimate for the relationship between the amount of pain relief at different amounts of oxytocin in the blood.

This is a study of participants that will receive an intravenous (IV) infusion of oxytocin (naturally occurring hormone that is made in the brain) with blood samples taken thereafter in order to create a formula to describe the concentrations of oxytocin in the blood over time (pharmacokinetics).

In this study healthy volunteers and people with knee arthritis so severe that there is a need for a joint replacement are recruited for a one day study. Each study participant will have 2 IV catheters placed (one in each arm). After placement of the IV catheters, 4 different levels of oxytocin will be given by IV infusion. Blood samples will be taken before the infusion begins and after each different level of the infusion. The blood will be drawn through the second IV catheter.

The study team will also do some tests to get a rough idea of how oxytocin changes perceptions on the skin and how this relates to the amount of oxytocin in the blood at the same time. The study team will study a painful perception by placing a probe on the skin and heating it to 113 degrees Fahrenheit for 5 minutes. Each study participant will score any pain that is experienced on a 0 to 10 scale.

DETAILED DESCRIPTION:
This is an unblinded, sequential study in which all participants will receive intravenous (IV) infusions of oxytocin in the same manner (except for safety reasons an adjustment at the highest level after review of the first 7 study participants as indicated in safety plan). In this study healthy people and with those with knee arthritis so severe that a joint replacement is needed are recruited for a one day study. Study participants will come to the Clinical Research Unit (CRU) and two IVs inserted; one in each forearm. Study participants will have an intravenous infusion of oxytocin at infusion rates that will result in a steady concentration of oxytocin in the blood for 15 minutes. The infusion rate will be increased every 15 minutes for a total of 4 targeted levels. Blood (5 millilitres (ml)) will be withdrawn through the IV not being used for infusion at the end of each of these infusion levels and the amount of oxytocin measured in the blood samples. This information will be analyzed by another group at Stanford University in the Pharmacokinetics/Pharmacodynamics (PK/PD) Core part of this application. The core group at Stanford University will use mathematics to test the accuracy of the infusion to target the blood concentration.

The main purpose of this study is to define the maximum effect oxytocin has on pain from a 5 minute heat probe applied to the skin and to get an estimate for the relationship between the amounts of pain relief at different amounts of oxytocin in the blood. The study team will use a commercially available device (Medoc TSA II) to heat a probe on the skin to 113 degrees Fahrenheit (45 degrees Celsius) for 5 minutes. Study participants will score any pain noted on a 0 to 10 scale, and most people find that pain rises during the 5 minutes, but remains mild, usually around only 1 or 2 on the 0 to 10 scale. The study team will do this 5 times during the study, once before the infusion and once during each of the 4 levels of infusion. From this the study team will calculate how the amount of oxytocin in the blood affects pain.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female > 18 and < 75 years of age, Body Mass Index (BMI) <40.
2. Generally in good health as determined by the Principal Investigator based on prior medical history, American Society of Anesthesiologists physical status 1, 2, or 3.
3. For healthy volunteers, normal blood pressure (systolic 90-140 mmHg; diastolic 50-90 mmHg) resting heart rate 45-100 beats per minute) without medication. For knee arthritis subjects, normal blood pressure or, for those with hypertension, pressure controlled with anti-hypertensives and with a resting heart rate 45-100 beats per minute.
4. Female subjects of child-bearing potential and those < 1 year post-menopausal, must be practicing highly effective methods of birth control such as hormonal methods (e.g., combined oral, implantable, injectable, or transdermal contraceptives), double barrier methods (e.g., condoms, sponge, diaphragm, or vaginal ring plus spermicidal jellies or cream), or total abstinence from heterosexual intercourse for a minimum of 1 full cycle before study drug administration.

Exclusion Criteria:

1. Hypersensitivity, allergy, or significant reaction to any ingredient of Pitocin®
2. Any disease, diagnosis, or condition (medical or surgical) that, in the opinion of the Principal Investigator, would place the subject at increased risk (active gynecologic disease in which increased tone would be detrimental e.g., uterine fibroids with ongoing bleeding), compromise the subject's compliance with study procedures, or compromise the quality of the data
3. Women who are pregnant (positive result for serum pregnancy test at screening visit), women who are currently nursing or lactating, women that have been pregnant within 2 years
4. Subjects with neuropathy, chronic pain, diabetes mellitus, or taking benzodiazepines or pain medications on a daily basis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Pharmacodynamics of heat pain after oxytocin | Baseline before any infusion 0 minutes
  Pain will be measured using a verbal Pain Scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to WORST PAIN IMAGINABLE.
Pharmacodynamics of heat pain oxytocin 16 pg/ml | Before Oxytocin infusion 15 minutes after baseline
  Pain will be measured using a verbal Pain Scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to WORST PAIN IMAGINABLE.
Pharmacodynamics of heat pain oxytocin 64 pg/ml | Before Oxytocin infusion 30 minutes after baseline
  Pain will be measured using a verbal Pain Scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to WORST PAIN IMAGINABLE.
Pharmacodynamics of heat pain oxytocin 256 pg/ml | Before Oxytocin infusion 45 minutes after baseline
  Pain will be measured using a verbal Pain Scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to WORST PAIN IMAGINABLE.
Pharmacodynamics of heat pain oxytocin 4pg/ml | After Oxytocin infusion 14 minutes after baseline
  Pain will be measured using a verbal Pain Scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to WORST PAIN IMAGINABLE.
Pharmacodynamics of heat pain oxytocin 16 pg/ml | After Oxytocin infusion 29 minutes after baseline
  Pain will be measured using a verbal Pain Scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to WORST PAIN IMAGINABLE.
Pharmacodynamics of heat pain oxytocin 64pg/ml | After Oxytocin infusion 44 minutes after baseline
  Pain will be measured using a verbal Pain Scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to WORST PAIN IMAGINABLE.
Pharmacodynamics of heat pain oxytocin 256 pg/ml | After Oxytocin infusion 59 minutes after baseline
  Pain will be measured using a verbal Pain Scale 0-10. 0 is equivalent to NO PAIN and 10 is equivalent to WORST PAIN IMAGINABLE.

SECONDARY OUTCOMES:
Pharmacokinetics of oxytocin in serum 4pg/ml | After Oxytocin infusion 15 minutes after baseline
  Blood will be sampled at the end of each infusion targeted to a set blood concentration of oxytocin. Serum will be separated, rapidly frozen, and later analyzed for oxytocin concentration. The accuracy of the pharmacokinetics will be assessed by difference between targeted and observed oxytocin concentrations.
Pharmacokinetics of oxytocin in serum 16 pg/ml | After Oxytocin infusion 30 minutes after baseline
  Blood will be sampled at the end of each infusion targeted to a set blood concentration of oxytocin. Serum will be separated, rapidly frozen, and later analyzed for oxytocin concentration. The accuracy of the pharmacokinetics will be assessed by difference between targeted and observed oxytocin concentrations.
Pharmacokinetics of oxytocin in serum 64pg/ml | After Oxytocin infusion 45 minutes after baseline
  Blood will be sampled at the end of each infusion targeted to a set blood concentration of oxytocin. Serum will be separated, rapidly frozen, and later analyzed for oxytocin concentration. The accuracy of the pharmacokinetics will be assessed by difference between targeted and observed oxytocin concentrations.
Pharmacokinetics of oxytocin in serum 256pg/ml | After Oxytocin infusion 60 minutes after baseline
  Blood will be sampled at the end of each infusion targeted to a set blood concentration of oxytocin. Serum will be separated, rapidly frozen, and later analyzed for oxytocin concentration. The accuracy of the pharmacokinetics will be assessed by difference between targeted and observed oxytocin concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: James C Eisenach, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No